CLINICAL TRIAL: NCT03521440
Title: Effects of Two Therapeutic Relaxation Programs on Health and Quality of Life Indicators of Elderly People Living in the Community
Brief Title: Therapeutic Relaxation, Health and Quality of Life
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Évora (Other)
Responsible Party: Principal Investigator, Gisela Cristina Resina Roque, Principal Investigator, University of Évora
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Universidade de Evora
Record Dates: First submitted 2018-04-20; First posted 2018-05-11 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Independent Living
Keywords: Therapeutic relaxation; Elderly; Community dwelling
MeSH Terms: interventions — Autogenic Training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Psychomotor Massage (Experimental): Participants will be randomly allocated to individual sessions, and will receive two 30-minute individual sessions per week, for 8 weeks.
  Interventions: Behavioral: Psychomotor Massage
- Progressive Muscle Relaxation (Experimental): Participants will participate in 30-minute group sessions, twice a week, for 8 weeks.
  Interventions: Behavioral: Progressive Muscle Relaxation
- Waiting List (No Intervention): Participants will maintain their daily routines through the experimental intervention period. After finishing all periods of data collection, participants will be invited to participate in one of the interventions previously offered to the experimental groups.

INTERVENTIONS:
Behavioral: Psychomotor Massage — Sessions will be conducted by a graduated therapist, experienced in Psychomotor Massage and weekly supervised by a specialist in this therapeutic approach. The Psychomotor Massage involves smoothly touching the head, upper and lower limbs, followed by micro-stretching and slow mobilisations of upper and lower limbs.
  Arms: Psychomotor Massage
Behavioral: Progressive Muscle Relaxation — Sessions will be conducted by a graduated therapist, experienced in Progressive Muscle Relaxation, and weekly supervised by a specialist in this therapeutic approach. The Progressive Muscle Relaxation protocol consists in tensing and releasing 16 muscle groups for several seconds, following a specific order.
  Other Names: Progressive Muscle Training
  Arms: Progressive Muscle Relaxation

SUMMARY:
Therapeutic relaxation has shown benefits for improving health and quality of life of community dwelling elderly people. Although little is known about the efficacy of a specific method of therapeutic relaxation - Psychomotor Massage - compared with other relaxation methods. Therefore, the present study aims to examine the effects of two therapeutic programs (Psychomotor Massage and Progressive Muscle Relaxation) on health and quality of life indicators of community dwelling elderly people. This randomized controlled trial will include an intervention period of 8 weeks for control and for the two experimental groups - attending 30-minute sessions, twice a week - and a follow-up period of 4 weeks without intervention. The evaluation will be performed 1) at baseline, 2) at post-intervention and pre-follow-up, and 3) at post-follow-up. The main study variables will be: daily activities, psychomotor abilities, cognitive functioning, emotional states, pain perception, quality of sleep, body awareness and body image, and quality of life. Health biomarkers will be also assessed through saliva analyses.

DETAILED DESCRIPTION:
According to World Health Organization, life expectancy of older people continues to rise, and by 2050, the proportion of the world's population above 60 years old will nearly double, from 12% to 22%. However, living longer does not mean living healthier. So, it is urgent to promote effective interventions in elderly people's health, quality of life and independency, aiming to be able to live autonomous in their homes and in community (WHO).

Aging involves changes on the body and its functions, for example the praxis skills, which leads to a visible decrease on the performance of Activities of Daily Living (ADL's) (e.g. self-care and domestic activities). These difficulties are also associated to dysfunctionality and poor quality of life. All of these decreases are also associated with emotional problems, sleep disorders, and pain.

In recent years, there has been a resurgence of interest in more integrative therapeutic interventions. In particular, therapeutic relaxation programs have been increasingly reported to be effective interventions for preventing the functional and emotional losses, associated to the aging process, as well as for promoting health and quality of life indicators. There is a specific method of therapeutic relaxation - Psychomotor Massage - that has been frequently applied in order to improve health and quality of life indicators of elderly people. However, to the best of the investigator's knowledge, no study has yet examined the effects of such innovative relaxation intervention method, particularly comparing them to the effects of a common therapeutic relaxation method, such as Progressive Muscle Relaxation.

Therefore, this experimental randomized controlled trial aims to examine the effects of two therapeutic interventions programs based on the relaxation techniques mentioned above in health and quality of life indicators (daily activities, psychomotor abilities, cognitive functioning, emotional states, pain perception, quality of sleep, body awareness and body image) of community dwelling Portuguese elderly people.

Subjects above 60 years living in the community will be invited to participate in this study and will be randomized by three groups: control, Psychomotor Massage, and Progressive Muscle Relaxation. Along the study, all patients will continue to receive the usual care from their medical providers. The study will include an intervention period of 8 weeks for control and for the two experimental groups - attending 30-minute sessions, twice a week - and a follow-up period of 4 weeks without intervention. Evaluation will be performed 1) at baseline, 2) at post-intervention and pre-follow-up, and 3) at post-follow-up. The study was approved by the Ethics Committee of the University of Évora, Portugal, and will be carried out in accordance with the standards set by the Declaration of Helsinki. The collected data will be fully encrypted to ensure the privacy of the participants.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 60 years
* Community dwelling
* Absence of cognitive impairment: cut-off < 22 at Mini Mental State Examination
* Able to participate at assessments
* Able to participate at therapeutic sessions

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2018-04-27 (Actual); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Activities of Daily Living (ADL's) | Change from baseline to 8 weeks, and change from baseline to 12 weeks
  The Portuguese version of Katz Index of ADL's grades (Duarte, Y. A. O., Andrade, C. L., & Lebrão, M. L., 2007) summarizes overall performance in six functions: bathing, dressing, going to toilet, transferring, continence and feeding. Time for application is 5 minutes. For each ADL the subject is classified as Dependent (0) or Independent (1). If the subject refuses, or is not used to a certain task, he is classified as Dependent in the respective activity. The final punctuation results from the sum of the 6 function scoring, and corresponds to the number of activities in which the subject is independent. The scale demonstrated adequate psychometric properties with strong reliability.
Psychomotor Skills | Change from baseline to 8 weeks, and change from baseline to 12 weeks
  The Portuguese version of Éxamen Géronto-Psychomoteur (P-EGP; Morais, Santos, & Lebre, 2017) is a measuring instrument of psychomotor skills of people above 60 years and aims to establish an individual psychomotor profile. The instrument consists of 17 items which assess: static and dynamic balance, joint mobilizations, praxis, fine motor skills of upper and lower limbs, knowledge of body parts, vigilance, perception, verbal and perceptive memory, spatial and temporal domain, and verbal and nonverbal communication. Each item is scored on a six-point scale, some with a set of sub-items inside. Time application is about 60 minutes. The P-EGP has been shown to have adequate psychometric properties.
Cognitive Functioning | Change from baseline to 8 weeks, and change from baseline to 12 weeks
  Wisconsin Card Sorting Test (WCST; Heaton, Chelune, Talley, Kay, & Curtiss, 1993) is constituted by carts that vary in term of their contents (forms, colours, figures). Subject is asked to correspond each answer-card to one of the four stimulus-card (on red triangle, two green stars, three yellow crosses, and four blue circles). WSCT implies the subject to develop a response pattern and implement an action plan, and provide ways to understand the cognitive flexibility, respond stiffness and problem-solving capacity. WSCT also involves the strategic planning, the organized visual processing, the processing speed, the skill to use environment feedback and select the relevant characteristics of stimuli, the work memory, impulsive response modulation, and the adoption of behaviours oriented to goals. The version that will be used has two blocks of 64 cards. Time application is about 15/30 minutes. The WCST shows good psychometric properties.
Humour and Emotional States | Change from baseline to 8 weeks, and change from baseline to 12 weeks
  The Portuguese version of short form Profile of Mood States (P-POMS; Viana, Almeida, & Santos, 2001) have 22 items, which allows to assess humour and emotional states. Respondents indicate in a 5-point likert scale (0=not at all to 4=extremely) to what extent each adjective describes them during the last week. Standard scoring of the POMS yields a global distress score and six subscales: Fatigue-Inertia, Vigour-Activity, Tension-Anxiety, Depression-Melancholy, Anger-Hostility, and Confusion-Disorientation. Completion of the POMS takes approximately 3 to 7 minutes (Viana et al., 2001). The Portuguese version of the POMS shows good psychometric properties (Viana et al., 2001).
Sleep Quality | Change from baseline to 8 weeks, and change from baseline to 12 weeks
  The Portuguese version of Pittsburgh Sleep Quality Index (P-PSQI; Del Rio João, Becker, Jesus, & Martins, 2017) is a 19-item questionnaire that measures sleep quality over the last month. The questionnaire comprises 19 items rated in a 3-point scale, that measures (1) subjective sleep quality, (2) sleep latency, (3) sleep duration, (4) habitual sleep efficiency, (5) sleep disturbances, (6) use of sleeping medication, and (7) daytime dysfunction. Higher scores indicate worst sleep quality. This questionnaire is easily understood and takes 5 to 10 minutes to be answered. The PSQI-PT has adequate psychometric properties.
Pain Perception | Change from baseline to 8 weeks, and change from baseline to 12 weeks
  The Portuguese version of Brief Pain Inventory - Short Form (P-BPI; Ferreira-Valente, Pais-Ribeiro, & Jensen, 2012) comprises 15 items which assess pain interference across seven ADL's (i.e. general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life) on 0 to 10 numerical scales. This version of the BPI retained the front and back body diagrams, the four pain severity items and seven pain interference items rated on 0-10 scales, and the question about percentage of pain relief by analgesics. This is a valid instrument, reproducible and sensible in detection, monitoring and characterization of pain, with excellent psychometric properties (Cronbach's alpha above .80).
Pain Perception | Change from baseline to 8 weeks, and change from baseline to 12 weeks
  The Visual Analogue Scale (VAS; Huskisson,1983) is a unidimensional self-rated instrument that allow quantify the subjective pain intensity. VAS is presented as a horizontal straight line of 10 centimetres, numbered from 0 (zero) to 10 (ten), which 0=without pain, 1 to 3=mild/light pain, 4 to 6=moderate pain, and 7 to 10=severe pain. This one is the worst pain possible. Participants are instructed to indicate a point on the line, correspondent to the intensity pain that they felt in the last week, including today. Standard is obtained through the measure between the point 0 (without pain) and the point marked by the participant. The score rate is from 0 to 10. VAS demonstrates good reliability scores through test-retest application with greater results with literate (r=.94, p<.001) compared with illiterate (r=.71, p=<.001).
Body Awareness and Dissociation | Change from baseline to 8 weeks, and change from baseline to 12 weeks
  The Portuguese version of Scale of Body Connection (P-SBC) is constituted by 2 subscales designed to assess body awareness and bodily dissociation in mind body intervention research, and 20 items self-report using a 5-point Likert scale format, in which 0=not at all; 1=a little bit; 2=some of the time; 3=most of the time; and, 4=all of the time. For scoring the Body Awareness (BA) subscale: sum score of items (items 1, 3, 4, 6, 8, 9, 12, 13, 14, 15, 17, 18) and divide by total number of items (12). For scoring the Body Dissociation (BD) subscale: sum score of items (items 2, 5, 7, 10, 11, 16, 19, 20) and divide by total number of items (8). For scoring Total Scale: revert the punctuation of the body dissociation subscale, sum the score of all items, and divide by total number of items (20).
  The P-SBC showed adequate psychometric properties (Cronbach's alpha coefficients of .86 for BA and .73 for BD).
Quality of Life | Change from baseline to 8 weeks, and change from baseline to 12 weeks
  The Portuguese version of Medical Outcomes Short-Form Health Survey (P-SF-36; Ferreira, 2000) is a non-specific questionnaire for health- related quality of life. The SF-36 consists of eight subscales as follows: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional and mental health. The P-SF-36 has been validated with adequate psychometric qualities.
Body Schema | Change from baseline to 8 weeks, and change from baseline to 12 weeks
  The evaluation of the body schema will be done through the Image Marking Procedure (Askevold, 1975). This procedure consists in a self-recording of certain body points (body height, acromio-clavicular joints, narrowest waist width and the trochanters of the femoral bones) on one piece of paper (1x1.5m) taped to the wall. The subjects are asked to stand in front of the paper and to imagine that they are looking at themselves through a mirror, while the investigator stands behind them and with his finger he touches the body points chosen for marking. The subjects are then asked to mark where they "see" these points in the "mirror". When the marking is finished, the investigator marks the correct position of the body points to compare these ones with the subjects' perceptive marks. This procedure shows good reliability, with values between 0.72 and 0.92.
Interoceptive Body Awareness | Change from baseline to 8 weeks, and change from baseline to 12 weeks
  The Portuguese translation of Multidimensional Assessment of Interoceptive Awareness (MAIA; Machorrinho, Veiga & Marmeleira (2017), will be used to measure interoceptive body awareness. This questionnaire has 32 items, which are organized in 8 different subscales (Noticing, Not-distracting, Not-worrying, Attention Regulation, Emotional Awareness, Self-Regulation, Body Listening and Trusting) and tested on a Likert scale, with six levels of ordinal response coded from 0 (never) to 5 (always). It was verified that the Portuguese version has good temporal reliability with correlation values of all scales between 0.52 and 0.83.
Corporal Appreciation | Change from baseline to 8 weeks, and change from baseline to 12 weeks
  The Body Assessment Scale (Avalos, Tylka e Wood-Barcalow, 2005) will be used in its translated and adapted version to the Portuguese language by Félix Neto (2011, quoted by Baldaia, 2013) to quantify the corporal appreciation. The Portuguese version consists of 14 items about the positive qualities of the body image and the answers are obtained on a Likert scale composed of 5 points from 1 (never) and 5 (always). Its reliability was verified by the application of Cronbach's alpha and the obtained value was α = 0.86 (Baldaia, 2013), which is similar with the results of both studies by Avalos, Tylka and Wood-Barcalow (2005) where the alpha values were equal to 0.91 and 0.93. Within this same subject, there will also be an open question about Body Image.

SECONDARY OUTCOMES:
Sleep Quality | Change from baseline to 8 weeks, and change from baseline to 12 weeks
  Patient will use the accelerometer ActiGraph wGT3X-BT during 4 days and 3 nights. Sleep Latency, Total Sleep Time, Wake After Sleep Onset and Sleep Efficiency will be assessed. The captures and records high resolution raw acceleration data, which is converted into a variety of objective activity and sleep measures using publicly available algorithms developed and validated by members of the academic research community. Available measures include: Body Position, Sleep Latency, Total Sleep Time, Wake After Sleep Onset, and Sleep Efficiency (ActiGraph, 2018).
Biochemical parameters (e.g., cortisol) | Change from baseline to week 4, change from week 4 to week 8, and change from week 8 to week 12
  Data (a saliva sample in a Salivette (r) tube) will be collect at: baseline, 10/15 minutes after baseline and immediately before the intervention and immediately after the intervention, at 1st, 8th, 16th sessions of therapeutic intervention. In follow-up assessment, data will be collect at baseline and 10/15 minutes after baseline, at 4th week. Samples will be collect at the same hour and period of the day in all moments of collection. After collected, were refrigerated. Therefore, participants of experimental groups will have 11 measurements, and participants of control group will have 8 measurements. Cortisol was measured in the standard unit of nmol/l.
Biochemical parameters (e.g., immunoglobulin A (sIgA)). | Change from baseline to week 4, change from week 4 to week 8, and change from week 8 to week 12
  Data (a saliva sample in a Salivette (r) tube) will be collect at: baseline, 10/15 minutes after baseline and immediately before the intervention and immediately after the intervention, at 1st, 8th, 16th sessions of therapeutic intervention. In follow-up assessment, data will be collect at baseline and 10/15 minutes after baseline, at 4th week. Samples will be collect at the same hour and period of the day in all moments of collection. After collected, were refrigerated. Therefore, participants of experimental groups will have 11 measurements, and participants of control group will have 8 measurements. sIgA concentration in the standard unit of µg/ml.
Biochemical parameters (e.g., a-amylase). | Change from baseline to week 4, change from week 4 to week 8, and change from week 8 to week 12
  Data (a saliva sample in a Salivette (r) tube) will be collect at: baseline, 10/15 minutes after baseline and immediately before the intervention and immediately after the intervention, at 1st, 8th, 16th sessions of therapeutic intervention. In follow-up assessment, data will be collect at baseline and 10/15 minutes after baseline, at 4th week. Samples will be collect at the same hour and period of the day in all moments of collection. After collected, were refrigerated. Therefore, participants of experimental groups will have 11 measurements, and participants of control group will have 8 measurements. Since most assay techniques employed to date make use of sAA's enzymatic activity, the most frequently used unit of measurement is enzyme units per milliliter (U/ml).
Biochemical parameters (e.g., C-reactive protein). | Change from baseline to week 4, change from week 4 to week 8, and change from week 8 to week 12
  Data (a saliva sample in a Salivette (r) tube) will be collect at: baseline, 10/15 minutes after baseline and immediately before the intervention and immediately after the intervention, at 1st, 8th, 16th sessions of therapeutic intervention. In follow-up assessment, data will be collect at baseline and 10/15 minutes after baseline, at 4th week. Samples will be collect at the same hour and period of the day in all moments of collection. After collected, were refrigerated. Therefore, participants of experimental groups will have 11 measurements, and participants of control group will have 8 measurements. C-reactive protein in the standard unit of mg/mL.

CONTACTS AND LOCATIONS:
Overall Officials: Catarina Pereira, PhD, Study Chair — University of Évora; Guida Veiga, PhD, Study Chair — University of Évora
Locations (1):
- Escola Superior de Enfermagem S. João de Deus, Evora, Portugal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] ActiGraph, L. (2018). ActiGraph wGT3X-BT. Retrieved April 10, 2018, from https://www.actigraphcorp.com/actigraph-wgt3x-bt/
- [Background] Askevold F. Measuring body image. Preliminary report on a new method. Psychother Psychosom. 1975;26(2):71-7. doi: 10.1159/000286913. PMID 1202548
- [Background] Avalos L, Tylka TL, Wood-Barcalow N. The Body Appreciation Scale: development and psychometric evaluation. Body Image. 2005 Sep;2(3):285-97. doi: 10.1016/j.bodyim.2005.06.002. Epub 2005 Aug 26. PMID 18089195
- [Background] Bair MJ, Wu J, Damush TM, Sutherland JM, Kroenke K. Association of depression and anxiety alone and in combination with chronic musculoskeletal pain in primary care patients. Psychosom Med. 2008 Oct;70(8):890-7. doi: 10.1097/PSY.0b013e318185c510. Epub 2008 Sep 16. PMID 18799425
- [Background] Baldaia, A. (2013). A atratividade física e o seu contributo para o envelhecimento bem-sucedido. Actas de Gerontologia, 1(1), 1-8.
- [Background] Cunha, L., & Mayrink, W. (2011). Influência da dor crônica na qualidade de vida em idosos. Revista Da Dor, 12(2), 120-124
- [Background] Del Rio Joao KA, Becker NB, de Neves Jesus S, Isabel Santos Martins R. Validation of the Portuguese version of the Pittsburgh Sleep Quality Index (PSQI-PT). Psychiatry Res. 2017 Jan;247:225-229. doi: 10.1016/j.psychres.2016.11.042. Epub 2016 Nov 28. PMID 27923147
- [Background] Ferreira-Valente, M. A., Pais-Ribeiro, J. L., & Jensen, M. P. (2012). Further Validation of a Portuguese Version of the Brief Pain Inventory Interference Scale. Clínica Y Salud, 23(1), 89-96. http://doi.org/10.5093/cl2012a6
- [Background] Ferreira PL. [Development of the Portuguese version of MOS SF-36. Part II --Validation tests]. Acta Med Port. 2000 May-Jun;13(3):119-27. Portuguese. PMID 11026151
- [Background] Gebretsadik M, Jayaprabhu S, Grossberg GT. Mood disorders in the elderly. Med Clin North Am. 2006 Sep;90(5):789-805. doi: 10.1016/j.mcna.2006.05.015. PMID 16962842
- [Background] Heaton, R., Chelune, G., Talley, J., Kay, G., & Curtiss, G. (1993). Wisconsin Card Sorting Test Manual: Revised and expanded. (Psychological Assessment Resources Inc, Ed.). Odessa.
- [Background] Huskisson, E. C. (1983). Visual Analogue Scales. In Raven Press (Ed.), Pain Measurement and Assessment (pp. 33-37). New York
- [Background] Lino VT, Pereira SR, Camacho LA, Ribeiro Filho ST, Buksman S. [Cross-cultural adaptation of the Independence in Activities of Daily Living Index (Katz Index)]. Cad Saude Publica. 2008 Jan;24(1):103-12. doi: 10.1590/s0102-311x2008000100010. Portuguese. PMID 18209838
- [Background] Machorrinho, J., Veiga, G., & Marmeleira, J. (2017). Propriedades psicométricas da versão portuguesa do Multidimentional Assessment of Interoceptive Awareness (MAIA). Universidade de Évora.
- [Background] Morais, A., Santos, S., & Lebre, P. (2016). Psychometric Properties of the Portuguese Version of the Éxamen Geronto-Psychomoteur (P- EGP). Educational Gerontology. http://doi.org/10.1080/03601277.2016.1165068
- [Background] Morais A, Santos S, Lebre P. Psychomotor, Functional, and Cognitive Profiles in Older People with and without Dementia:What Connections? Dementia (London). 2019 May;18(4):1538-1553. doi: 10.1177/1471301217719624. Epub 2017 Jul 28. PMID 28752771
- [Background] Neves, C. F., Price, C. J., & Carvalheira, A. (2017). The psychometric properties of the Scale of Body Connection (SBC) in a Portuguese sample. Psychology, Community & Health, 6(1), 158-169. http://doi.org/10.5964/pch.v6i1.223
- [Background] Orsal O, Alparslan GB, Ozkaraman A, Sonmez N. The effect of relaxation exercises on quality of sleep among the elderly: holistic nursing practice review copy. Holist Nurs Pract. 2014 Jul-Aug;28(4):265-74. doi: 10.1097/HNP.0000000000000032. PMID 24919097
- [Background] Rubenstein LZ. Falls in older people: epidemiology, risk factors and strategies for prevention. Age Ageing. 2006 Sep;35 Suppl 2:ii37-ii41. doi: 10.1093/ageing/afl084. PMID 16926202
- [Background] Santana I, Duro D, Lemos R, Costa V, Pereira M, Simoes MR, Freitas S. [Mini-Mental State Examination: Screening and Diagnosis of Cognitive Decline, Using New Normative Data]. Acta Med Port. 2016 Apr;29(4):240-8. doi: 10.20344/amp.6889. Epub 2016 Apr 29. Portuguese. PMID 27349775
- [Background] Seidler RD, Bernard JA, Burutolu TB, Fling BW, Gordon MT, Gwin JT, Kwak Y, Lipps DB. Motor control and aging: links to age-related brain structural, functional, and biochemical effects. Neurosci Biobehav Rev. 2010 Apr;34(5):721-33. doi: 10.1016/j.neubiorev.2009.10.005. Epub 2009 Oct 20. PMID 19850077
- [Background] Tel, H. (2013). Sleep quality and quality of life among the elderly people. Neurology Psychiatry and Brain Research, 19(1), 48-52. http://doi.org/10.1016/j.npbr.2012.10.002
- [Background] Viana, M. F., Almeida, P. L. de, & Santos, R. C. (2001). Adaptação portuguesa da versão reduzida do Perfil de Estados de Humor - POMS. Análise Psicológica, 1(19), 77-92. Retrieved from http://publicacoes.ispa.pt/index.php/ap/article/view/345
- [Background] World Health Organization. (2017). Mental health of older adults. Retrieved from http://www.who.int/mediacentre/factsheets/fs381/en/